CLINICAL TRIAL: NCT00112216
Title: Specific Immunotherapy of Skin Melanoma Patients With Antigenic Peptides and Immunological Analysis of the Vaccine Site Sentinel Lymph Node
Brief Title: Immunotherapy of Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Ralph Venhaus, MD, Head of Clinical and Regulatory Affairs, Ludwig Institute for Cancer Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD 1998-009
Record Dates: First submitted 2005-05-31; First posted 2005-06-01 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2009-03

CONDITIONS: Melanoma
Keywords: Immunotherapy; Vaccination; Melanoma; Melan-A/Mart-1 peptide; Flu peptide; Mage-A10 peptide; SB AS-2 adjuvant; Montanide adjuvant
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Melan-A analog peptide
Biological: FluMa peptide
Biological: Mage-A10 peptide
Biological: SB AS-2 adjuvant
Biological: Montanide adjuvant

SUMMARY:
The purpose of this study is to test whether vaccination with antigenic peptides induces an immune response in the vaccine site sentinel lymph node of patients with microscopically detectable lymph node melanoma metastases.

DETAILED DESCRIPTION:
The study is designed for patients with skin melanoma and lymph node micrometastasis previously diagnosed by a sentinel node procedure. As a result of their diagnosis, the patients are scheduled for lymph node dissection. Before this is done, patients are vaccinated with antigenic peptides. The peptides are mixed with the adjuvant SB AS-2 or Montanide and injected in a lower limb not affected by the disease. The skin site of vaccine injection is marked with a permanent pen where, two weeks later, patent blue and 99technetium is injected. These markers allow one to locate the vaccine site sentinel node (VSSN) which will be removed during the lymph node dissection at the diseased limb.

The aim of the study is to test whether the vaccine has induced an immune response in the lymph node that drains the vaccine site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with microscopically detectable lymph node metastases
* Positive detection of the Melan-A gene +/- MAGE-10 in positive sentinel node or primary tumor tissue by polymerase chain reaction (PCR) analysis of mRNA and/or by immunohistochemistry using monoclonal antibodies
* Human leukocyte antigen-A2 (HLA-A2) positive

Exclusion Criteria:

* Previous splenectomy or radiotherapy to the spleen
* Treatment with systemic antihistamines, corticosteroids, or non-steroidal anti-inflammatory drugs (except occasional or low dose non-steroidal anti-inflammatory drugs such as 100 mg aspirin/day) within 4 weeks of entry into the study
* Heart disease (New York Heart Association [NYHA] Class III or IV)
* Serious illness, e.g. active infections requiring antibiotics, bleeding disorders or other diseases considered by the investigator to have potential for interfering with obtaining accurate results from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1999-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Melan-A, Flu and Mage specific CD8+ T-cell reactivity obtained from different body sites (vaccine site draining lymph node, other lymph node) will be measured by Tetramers and Elispot assays

SECONDARY OUTCOMES:
Safety and toxicity of antigenic peptides administered with high dose adjuvant will be assessed according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Speiser, MD, Principal Investigator — Ludwig Institute for Cancer Research
Locations (1):
- Ludwig Institute for Cancer Research + Multidisciplinary Oncology Center at the Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Ayyoub M, Zippelius A, Pittet MJ, Rimoldi D, Valmori D, Cerottini JC, Romero P, Lejeune F, Lienard D, Speiser DE. Activation of human melanoma reactive CD8+ T cells by vaccination with an immunogenic peptide analog derived from Melan-A/melanoma antigen recognized by T cells-1. Clin Cancer Res. 2003 Feb;9(2):669-77. PMID 12576434